CLINICAL TRIAL: NCT00091806
Title: An Open-Label, Clinical Trial Evaluating the Safety and Pharmacokinetics of Two Dose Schedules of Panitumumab in Subjects With Advanced Solid Tumors
Brief Title: Two Dose Schedules of Panitumumab in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20030251
Record Dates: First submitted 2004-09-17; First posted 2004-09-21 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Tumors; Oncology; Solid Tumors
Keywords: Targeted Therapy; Solid tumors; ABX-EGF, panitumumab; EGFr; Immunex, Abgenix, Amgen; Monoclonal Antibody
MeSH Terms: conditions — Neoplasms | interventions — Panitumumab

ARMS (2):
- Cohort 1 (Experimental): 6mg/kg of panitumumab administered once every 2 weeks until subjects develop disease progression or are unable to tolerate the study drug
  Interventions: Drug: panitumumab (ABX-EGF)
- Cohort 2 (Experimental): Panitumumab 9 mg/kg administered once every 3 weeks until subjects develop disease progression or are unable to tolerate the study drug.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: panitumumab (ABX-EGF) — 6 mg/kg once every 2 weeks
  Arms: Cohort 1
Drug: Panitumumab — 9 mg/kg once every 3 weeks
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of two dose schedules of panitumumab in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of advanced solid tumors that are refractory to at least 1 standard therapy or for which no standard therapy is available and have not received more than 3 prior treatment regimens (not inclusive of hormonal therapies for breast and prostate cancer subjects) for the advanced solid tumor (tumor must be diagnosed by standard criteria for the specific tumor type)
* Measurable disease or evaluable (non-measurable) disease per RECIST guidelines (all sites of disease must be evaluated within 28 days before enrollment)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of > 3 months as documented by the investigator
* If history of other primary cancer, subject will be eligible only if she or he has:

  * Non-melanomatous skin cancer, not requiring treatment
  * Curatively treated cervical carcinoma in situ
  * Other primary solid tumor curatively treated with no known active disease present for the last 5 years and no treatment administered for the last 3 years
* Man or woman 18 years of age or older
* Paraffin-embedded tumor tissue (from primary or metastatic tumor tissue) available for immunohistochemistry studies of EGFr expression (biopsy or archived tissue are acceptable). The immunohistochemical EGFr staining and evaluation must be conducted at the designated central laboratory using the DakoCytomation EGFR pharmDXTM kit. Local laboratory EGFr expression is not permitted for the purpose of eligibility in this study
* Hematologic function, as follows:

  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * Hemoglobin > 8 g/dL
* Renal function, as follows:

  o Creatinine < 2.0 mg/dL
* Hepatic function, as follows:

  * Aspartate aminotransferase (AST) < 3 x ULN (if liver metastases ≤ 5 x ULN)
  * Alanine aminotransferase (ALT) < 3 x ULN (if liver metastases ≤ 5 x ULN)
  * Bilirubin < 2 x ULN
* Competent to comprehend, sign, and date an IEC/IRB-approved informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-08; Primary Completion 2006-04 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and PK of 2 dose schedules of panitumumab in subjects with advanced solid tumors, refractory to or with no available standard therapy. | 2 years

SECONDARY OUTCOMES:
To asses the immunogenicity and efficacy of 2 dose schedules of panitumumab in subjects with advanced solid tumors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Stephenson JJ, Gregory C, Burris H, Larson T, Verma U, Cohn A, Crawford J, Cohen RB, Martin J, Lum P, Yang X, Amado RG. An open-label clinical trial evaluating safety and pharmacokinetics of two dosing schedules of panitumumab in patients with solid tumors. Clin Colorectal Cancer. 2009 Jan;8(1):29-37. doi: 10.3816/CCC.2009.n.005. PMID 19203894
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20030251.pdf
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/